CLINICAL TRIAL: NCT06498414
Title: SSTARLET: Shorter and Safer Treatment Regimens for Latent TB
Brief Title: Shorter and Safer Treatment Regimens for Latent TB
Acronym: SSTARLET
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Dick Menzies, Senior Investigator at Research Institute of McGill University Health Center, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OCT-194228
Record Dates: First submitted 2024-04-29; First posted 2024-07-12 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-06

CONDITIONS: Tuberculosis Infection, Latent
Keywords: Tuberculosis infection; Rifampin; Short treatment for latent tuberculosis; High dose rifampin
MeSH Terms: conditions — Latent Tuberculosis | interventions — Levofloxacin; rifapentine

STUDY DESIGN:
Intervention Model Description: We plan an initial randomization ratio of 1:2:2 for 4 months of rifampin 10mg/kg (4R10), 2 months of rifampin 20mg/kg (2R20), and one month levofloxacin and rifapentine (1LP).
Who Masked: Outcomes Assessor
Masking Description: Outcomes (Adverse event and tuberculosis (TB) disease) judge by independent blinded panel
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 4 months standard dose rifampin (4R10) (Active Comparator): 120 doses daily self-administered rifampin at 10 mg/kg/day (max. 600 mg/day)
  Interventions: Drug: rifampin standard arm
- 2 months high dose rifampin (2R20) (Experimental): 60 doses daily self-administered rifampin at 20 mg/kg/day (max.1200 mg/day)
  Interventions: Drug: rifampin double dose
- 1 month levofloxacin and rifapentine (1LP) (Experimental): 30 doses daily self-administered levofloxacin (15 mg/kg/day, max. 750 mg/day and rifapentine (10mg/kg/day, max. 600mg)
  Interventions: Drug: levofloxacin and rifapentine

INTERVENTIONS:
Drug: rifampin standard arm — 120 doses daily self-administered rifampin at 10mg/kg/day (max 600mg/day)
  Other Names: 4R10
  Arms: 4 months standard dose rifampin (4R10)
Drug: rifampin double dose — 60 doses daily self-administered rifampin at 20 mg/kg (max. 1200 mg/day)
  Other Names: 2R20
  Arms: 2 months high dose rifampin (2R20)
Drug: levofloxacin and rifapentine — 30 doses daily self-administered levofloxacin (15 mg/kg, max 750mg/day and rifapentine (10mg/kg, max: 600mg)
  Other Names: 1LP
  Arms: 1 month levofloxacin and rifapentine (1LP)

SUMMARY:
Our study rationale is based on:

1. Tuberculosis Preventive Treatment (TPT) is given to healthy people and needs to be safe;
2. Tuberculosis Preventive Treatment (TPT) with shorter regimens are superior with respect to acceptance, completion, and costs;
3. 4 months of Rifampin 10mg/kg (4R10) is the safest regimen, but is completed by <80% of patients;
4. The safety of 2 months of Rifampin 20mg/kg (2R20) is similar to that of 4 months of Rifampin 10mg/kg (4R10), but completion is a concern;
5. 1-month regimens have promising efficacy;
6. Safety and tolerability must be carefully assessed with comparisons to 4 months of Rifampin 10mg/kg (4R10), and head-to-head with each other.

OBJECTIVES: The investigator will use a Bayesian adaptive Phase 2 randomized open-label trial design to test at least three experimental Tuberculosis Preventive Treatment (TPT) regimens to identify at least one regimen of ≤2 months duration that has non-inferior safety, completion, and tolerability in adults and children relative to the reference Tuberculosis Preventive Treatment (TPT) regimen. The shortest, safest, and best tolerated regimen identified in this Phase 2 trial will be tested for effectiveness and efficacy in a Phase 3 trial.

Specific Tuberculosis Preventive Treatment (TPT) regimens (All are daily and self-administered) Reference: Rifampin at a dose of 10 mg/kg/day for 4 months (4R10); Experimental: 1) Rifampin at 20 mg/kg/day for 2 months (2R20); (2) one month Levofloxacin and Rifapentine (1LP). At a later stage a 3rd experimental regimen will be selected and added: one another novel 1-2-month regimen identified from pre-clinical and clinical studies. When selected, this will be explained fully including preliminary data on safety and efficacy in an amended protocol and consent - which will be submitted for ethics and regulatory approval at that time).

DETAILED DESCRIPTION:
DESIGN: The investigator proposes to assess safety, completion, and tolerability of three experimental Tuberculosis Preventive Treatment (TPT) regimens in an open label multi-arm Phase 2 adaptive trial. The investigator will start the trial with the reference 4 months of Rifampin 10mg/kg (4R10) and first two experimental regimens (2 months of Rifampin 20mg/kg (2R20), one month Levofloxacin and Rifapentine (1LP); if either experimental regimen does not meet pre-determined selection criteria, the experimental regimen will be dropped; if acceptable, enrolment will be reduced so that a 3rd new experimental regimen may be tested. This will be either one month of Isoniazid plus rifapentine (1HP), or an entirely novel regimen; this choice will be made on the basis of all available pre-clinical evidence and clinical studies. Note that when this 3rd regimen is selected the protocol and informed consent will be revised to include a description of this regimen, including results from all pre-clinical and clinical studies of efficacy, tolerability and safety. The revised consent and protocol will be submitted, as an amendment, for ethics and regulatory review. The available pre-clinical evidence will include ongoing work by one of the Principal Applicant and co-Aplicant and clinical studies. Randomization will be adjusted as regimens are added or dropped. Including new regimens, and dropping those with unacceptable safety, completion, and/or tolerability, will improve trial efficiency and timeliness of results. Regimens will be assessed for acceptability (qualitatively), health system and patient costs, and drug exposure (based on pharmacokinetics (PK)) to understand potential trade-offs between dose, duration, acceptability, tolerability, and costs. After the first 100 persons have completed treatment for each new Tuberculosis Preventive Treatment (TPT) regimen, the investigators plan an early safety analysis to identify whether a regimen has substantially higher rates of severe Adverse Event (AE); if this were to occur, enrolment to that arm will stop. After 400 participants have completed each of the two initial experimental regimens, the investigators plan an 'Initial regimen selection analysis. Regimens will continue enrolment if the regimen meet the criteria for non-inferior safety, completion, and tolerability compared to that of 4 months of Rifampin 10mg/kg (4R10). Margins for non-inferiority are stricter for safety - our primary outcome -than for completion and tolerability, our secondary outcomes (see section 2.10 for non-inferiority margins and justification). The investigators have planned for 24 months of enrolment to evaluate at least three experimental regimens. Enrolment will stop after 400 persons have been enrolled to experimental regimen 3; the Final regimen selection analysis will determine which regimen will continue in a Phase 3 trial.

STUDY SITES: Calgary, Edmonton, Montreal, Ottawa, Toronto, Vancouver, and Winnipeg (Canada); Cotonou (Benin); Manaus (Brazil); Bandung (Indonesia); and Ho Chi Minh City (Vietnam).

PLANNED ENROLMENT: The investigator plans to enroll a total of 1800 participants. Enrolment will continue at all sites until this number is reached, then enrolment will stop at all sites at the same time. In other words, there is no fixed maximum target enrolment for each site; rather, this is a cooperative trial in which all sites strive to achieve together the required enrolment. The first 'regimen selection analysis' will be conducted after 400 participants have completed treatment in each experimental arm. The investigators anticipate enrolling 700 total participants in 13-14 months on the basis of our past performance at all sites and adding three new sites in Canada, plus Brazil, and Benin, which were high enrolling sites in our 4v9 trial. After participant 700 has been enrolled, the 3rd experimental regimen will be added, and randomization will be modified so that equal numbers are allocated to the 3rd regimen, and to all continuing regimens (i.e., a ratio of 3:1:1:1 for 3rd experimental: 4 months of Rifampin 10mg/kg (4R10), 2 months of Rifampin 20mg/kg (2R20), and one month levofloxacin and rifapentine (1LP), until the first regimen selection analysis is complete. To ensure timely initiation, this 3rd regimen must be selected by the end of Year 1 (at the latest), so that ethics and regulatory approval can be obtained for all sites. After the first regimen selection analysis is complete, enrolment to experimental regimens 1 and/or 2 may stop. The investigators expect 1800 total enrollees by mid-Year 3, providing 400 enrollees to the 3rd experimental regimen and an added 400 to be split between 4 months of Rifampin 10mg/kg (4R10) and experimental regimens 1 and/or 2.

RANDOMIZATION: Randomization will be by computer-generated random sequences, in blocks of variable size, and stratified by site to account for previously observed differences between sites in rates of completion and Adverse Events (AEs). The investigator will allocate all members of the same household (for household contacts), to the same arm. The randomization program will be developed by the same group as for our prior Research Clinical Trials (RCTs) (demo: https://2r2-demo-ltb.cred.ca Identification: 2r2-demo Password: 2R2-demo123456789!). This will verify eligibility and if another household member was randomized. The investigator plan an initial randomization ratio of 1:2:2 for 4 months of Rifampin (4R10), 2 months of Rifampin (2R20), and 1 month Levofloxacin and Rifapentine (1LP); fewer participants need to be randomized to the 4 months of Rifampin (4R10) arm given the availability of results from our three prior 4 months of Rifampin (4R10) trials at the same sites, with the same inclusion/exclusion criteria, similar participant characteristics, and very consistent rates of Adverse Event (AE) and completion DURATION OF TREATMENT AND FOLLOW-UP: The investigators wish to ensure that burden on participants of in-person follow-up visits is similar in all arms, reduce effects of differential follow-up on treatment completion, and also reflect usual care follow-up procedures for the standard arm. Given the well-established safety of 4 months rifampin (4R), most patients receiving this regimen outside of a study (ie routine care) are seen in-person only once after 4 weeks of treatment and are called by telephone every month thereafter. Hence persons randomized to 4 months of Rifampin 10mg/kg (4R10) will be seen at 2 weeks, called by telephone at 4, 8, and 12-13 weeks, then come for a final end-of-treatment in person visit. Those randomized to one month levofloxacin and rifapentine (1LP) will be seen for routine follow-up visits at 2 weeks of treatment and end-of-treatment (4 weeks). Persons randomized to 2 months of Rifampin 20mg/kg (2R20) will be seen in person at 2 weeks, and end-of-treatment (8-9 weeks). To allow detection and response to poor tolerability, participants in both experimental arms will be called evaluated at 2 weeks; if symptoms of intolerability are reported and if judged not an adverse event, the participant will be offered the opportunity to switch to 4 months of Rifampin 10mg/kg (4R10). Routine blood tests (complete blood count, alanine transaminase (ALT), bilirubin) and blood sampling for population pharmacokinetics (PK) will be performed at 2 weeks for all persons. For all regimens, participants will be called 2 weeks after the last dose taken to detect possible late Adverse Events (AEs). During each in-person visit, participants will complete an interviewer-administered symptom questionnaire, pill counts will be performed, and new pills dispensed. During telephone follow-up visits, the same symptom questionnaire will be administered, and participants asked to report pills remaining. If a participant wishes to stop therapy, the benefits of Tuberculosis Preventive Treatment (TPT) will be re-emphasized, but the participant may stop without negative consequences. To reduce bias due to differential efforts to enhance adherence, staff will follow Standard Operating Procedures (SOPs) written pre-trial.

In summary, safety monitoring will be the most intensive for persons allocated to one month levofloxacin and rifapentine (1LP), for which the investigator have the least safety data, still quite intensive monitoring for persons allocated to 2 month rifampin (2R20), for which the investigator have reassuring safety data from approximately 450 participants, and much less monitoring for the standard regimen, but which aligned with current practice. In addition to routine visits and calls, participants will also be encouraged to call the study coordinator (the study participant will be given the study cell phone number which is carried by study personnel 24/7), or TB clinic nurses at any time if the participant experience symptoms or other problems, the participant think might be related to the study medications. The participant will also be encouraged to come as 'walk-ins' to the clinic at any time if symptoms or concerns arise.

Post-treatment follow-up to detect incident tuberculosis (TB) disease: Participants will be contacted every 3 months until 26 months post-randomization and asked about current symptoms of active tuberculosis (TB), any intercurrent diagnoses of active tuberculosis (TB), or hospitalization for any reason. Suspected active tuberculosis (TB) will be investigated. At study end, the investigators will also cross-check all participants with local nominal registries of tuberculosis (TB) disease notifications to detect other participants diagnosed with tuberculosis (TB) disease.

PLANNED ANALYSES: Safety: Our primary analysis is performed within the Bayesian framework using a beta-binomial model that places a non-informative (flat) prior distribution on the rate parameter. Statistical significance is defined with respect to the posterior probability of non-inferiority. The investigators will use robust dynamic borrowing methods to incorporate the prior trial data available on the reference treatment into the analysis. The weight assigned to previous data will be determined in a sensitivity analysis to ensure controlling the type I error. Secondary analyses will include a Bayesian generalized mixed effect model to account for clustering.

Regimen completion and tolerability: The investigators will use the same beta-binomial model for these two secondary outcomes. For both outcomes, the investigators specify a larger non-inferiority margin of 10% as the maximum tolerated difference, and a more permissive probability threshold of 90% for concluding non-inferiority. This means an experimental treatment will be deemed non-inferior to 4R10 with respect to either tolerability or completion if the posterior probability of non-inferiority exceeds 90%.

Acceptability: Transcribed, translated, and anonymized interview recordings will be thematically analyzed, drawing on acceptability frameworks, to elucidate participant-prioritized criteria for Tuberculosis Preventive Treatment (TPT) acceptability. The investigators will use researcher reflexivity, inter-rater reliability, contextualization, and gather thick descriptions to enhance rigor. Qualitative findings will contextualize quantitative results, be triangulated to inform treatment tolerability and adherence data, and guide knowledge translation activities.

TB Disease: This Phase 2 trial is underpowered for this outcome. Hence, the investigators will describe the incidence of TB disease by arm, using total person-time of follow-up of the modified intention to treat (MITT) population.

INTERIM SAFETY ANALYSES: To optimize the safety of study participants and identify any major excess in Adverse Event (AE) rates, the investigators plan safety analyses after the first 100 participants are randomized to each new regimen. The data and safety monitoring board (DSMB) will be blinded to study arm during review. If needed, unblinding will be done. The data and safety monitoring board (DSMB) will "make judgments about the strength of the evidence and the absolute magnitude and seriousness of any safety signals", rather than absolute 'stopping rules'.

PLANNED SUB-GROUP ANALYSES: The investigators will examine the association of severe Adverse Events (AEs) with age, sex, country, and comorbidities, and completion and tolerability by age, sex, country, and indication for Tuberculosis Preventive Treatment (TPT).

ELIGIBILITY:
Inclusion Criteria:

* Adults, and children aged ≥5 years with weight of > 15Kg.
* Positive test for TB infection: either Tuberculin test (>5mm, or >10mm, based on epidemiologic and clinical factors and interpreted following local guidelines) or interferon gamma release assay based on Manufacturer's criteria; and,
* Recommended for Tuberculosis Preventive Treatment (TPT), following Canadian guidelines (for Canadian sites), and World Health Organization (WHO) guidelines (for international sites).

Exclusion Criteria:

* Current tuberculosis (TB) disease - detected pre-enrolment with symptom screen, chest x-ray, and confirmatory microbiological (culture or genotypic) testing as needed; Prior to referral to research staff (research clinic) for consideration as potential participants, all persons must undergo symptoms screen and a chest Xray. If chest Xray is not available, then a negative results from a GeneXpert MTb RIF Ultra of spontaneous (expectorated) sputum will be considered sufficient to exclude TB disease pre-referral. If Chest Xray is abnormal or symptoms consistent with TB disease are present then at least two AFB smears and mycobacterial cultures must be done, and must be negative, or one GeneXpert MTb Rif Ultra must be negative before enrolment
* Children aged 0-4 years;
* Persons weighing <15 kg.
* Women who are pregnant or breast-feeding;
* Women of child-bearing potential and not willing to take an effective form of contraception (non-hormonal) during the treatment phase;
* Documented prior treatment for tuberculosis (TB) infection or disease;
* Pre-enrolment - alanine transaminase (ALT), White Blood Cells, platelets or hemoglobin that correspond to a Grade 3 adverse event (AE);
* Rifampin or rifapentine contra-indicated - due to allergy/hypersensitivity to any rifamycin (rifampin, rifabutin or rifapentine), or, drug interactions too difficult to manage;
* Have a prolonged QT interval on routine ECG pre-enrolment or take any medications that may prolong the QT interval and that are not recommended to take with a fluroquinolone. (See APPENDIX 5 in supplement for list of medications contra-indicated to take with Levofloxacin);
* Household contacts (HHC) of index TB patients with phenotypic or genotypic resistance to Rifampin or Levofloxacin. HHC may be enrolled, then excluded post-randomization, if resistance is identified later. Note that all sites routinely test Rifampin resistance in all people newly diagnosed to have TB disease, but do not test routinely for susceptibility to Levofloxacin unless Rifampin resistance is detected. Hence HHCs may be enrolled if their Index TB patient is Rifampin susceptible, even if Drug Susceptibility Testing to Levofloxacin is not done and/or not available.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1800 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Severe treatment-related Adverse Events (AE) | From the start of the treatment until 2 weeks after the treatment completion
  The investigators wish to capture all clinically relevant Adverse Event (AEs) defined as events that are possibly or probably treatment-related and result in death, hospitalization, or investigators' decision to discontinue study drug. These are defined as Grade 3-5 Adverse Event (AEs) of any type, plus Grade 1-2 rash/allergy. Because allergic reactions that are often detected by participants at an early stage carry the risk of progressing to more advanced manifestations if therapy is continued, stopping study drug is mandated with any Grade allergic reaction. If a suspected treatment-related Adverse Event (AE), or any hospitalization or death occurs during treatment phase (up to 2 weeks after the last dose of study drug taken), the site will file initial and final Adverse Event (AE) reports that will be sent for adjudication by the Adverse Event (AE) panel who will be blinded to study arm.

SECONDARY OUTCOMES:
Completion | at the end of the treatment (1 month, 2 months or 4 months)
  Completion will be defined as taking at least 80% of prescribed doses within 150% of allowed time. This outcome will be based on the number of pills dispensed and counted during treatment follow-up visits, along with time from randomization until the date that ≥80% of doses of study drug are taken. This threshold is derived from a large-scale trial in which efficacy was significantly greater in persons who took at least 80% of doses.
Tuberculosis Preventive Treatment (TPT)-related symptoms - Tolerability | 2 weeks after the treatment has started in all arms
  The investigators found that reporting symptoms at the time of routine treatment phase follow-up visits, which the patient's provider did not consider an AE and so did not discontinue treatment, occurred significantly more frequently with 2 months of Rifampin 30mg/kg (2R30) than 2 months of Rifampin 20mg/kg (2R20) or 4 months of Rifampin 10mg/kg (4R10); this was associated with subsequent patient decision to stop Tuberculosis Preventive Treatment (TPT) in our 2R2 trial and our 4v9 trial. Thus, symptoms will be captured with a questionnaire, assessing the 10 most commonly reported symptoms at the time of routine follow-up visits in these previous trials.
Patient preferences and acceptability of Tuberculosis Preventive Treatment (TPT) | 2 weeks after the treatment has started in all arms
  The impacts of different Tuberculosis Preventive Treatment (TPT) regimens on adherence, quality of life, and perceived trade-offs between pill burden, tolerability, and duration will be explored using qualitative methods informed by treatment acceptability frameworks, including those used in discrete choice experiments and the evaluation of broader disease prevention interventions. A purposive sample will include approximately 10 participants per arm in each country, with equal representation from men and women, key affected populations in each country, and participants who completed or decided to stop early. For pediatric participants we will interview their adult caregivers. They will be recruited for two private semi-structured, audio-recorded interviews. The first interview (10-15 min), after two weeks of treatment, will inquire on first impressions of treatment, including tolerability, impact on daily life, and early adherence issues.
Plasma drug exposures | 2 weeks after the treatment has started in all arms
  Pharmacokinetics (PK) of rifampin, levofloxacin, and rifapentine will be assessed after two weeks of therapy in all arms. An intensive Pharmacokinetics (PK) sub-study will be performed at sites with facilities and trained personnel to characterize peak concentrations (Cmax) and total drug exposures over the dosing interval (AUC). Serial venous blood samples will be collected at 0, 0.5, 1, 2, 4, 8, and 12 h after drug intake in 10 participants per sub-group in younger children aged 5-9 years, in adults, and also in people living with HIV on antiretroviral (30 total per arm). A population PK sub-study (e.g., either at 1, or 2, or 3, or 4, or 6 h after drug intake) will also be performed in consenting participants at all sites to assess determinants of Pharmacokinetics (PK) variability and the association of drug exposure on study outcomes.
  A separate sub-study in breastfeeding women will be performed to assess PK profiles of a single dose of RIF, LFX, INH, RPT, and BDQ (PRiMe study).
Assess both health system and patient/family costs | 2 weeks after the treatment has started in all arms
  The investigators will assess both health system and patient/family costs using a bottom-up micro-costing approach and patient questionnaires. The investigators will perform activity-based costing informed by all relevant health services used by participants including visits, medications, tests, and hospitalizations (all collected in study case report forms (CRFs), and cost these items based on previous work. To estimate patient/family costs during treatment phase, the investigators will administer a questionnaire that we have used previously about out-of-pocket costs (e.g., transport, food) and time taken for Tuberculosis Preventive Treatment (TPT) related activities; this will be assessed in 20 participants per country and study arm. For employed persons, the investigators will value indirect costs of time using the mean wage in their jurisdiction (province or country) for their job title; for unemployed persons, the investigators will use the mean wage in the same jurisdiction.
Active TB is suspected within 26 months of randomization | From start of the treatment until 26 months after the randomization
  If active TB is suspected within 26 months of randomization, this will be investigated, managed, and reported in accordance with detailed standard operating procedures (SOPs). The final diagnosis will be based on microbiological confirmation. If not confirmed, the diagnosis will be based on the judgement of probable tuberculosis (TB) disease by the majority of a blinded 3-member independent panel that will review clinical information, microbiologic and radiologic results, and treatment response.

CONTACTS AND LOCATIONS:
Overall Officials: Dick Menzies, MD, Principal Investigator — RI-MUHC
Locations (13):
- Centre National Hospitalier Universitaire de Pneumo Phtisiologie de Cotonou (CNHU-PPC), Cotonou, Benin
- Manaus, Manaus, Brazil
- Canada (9):
  - Unviversity of Calgary, Calgary, Alberta
  - The Governors of the University of Alberta, Edmonton, Alberta
  - BCCDC TB clinic, Vancouver, British Columbia
  - University of Manitoba, Winnipeg, Manitoba
  - University of Ottawa, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - MUHC, Montreal, Quebec
  - Hopital du Sacré-Coeur de Montreal, Montreal, Quebec
- Universitas Padjadjaran, Klinik Penelitian Tuberculosis (TB research clinic), Bandung, Indonesia
- Vietnam, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Protocol and consent form will be available for data sharing once approved by research ethical review board. A detailed plan for data sharing of other study documents and/or data is under definition and will be posted during the trial.
Supporting Information: Study Protocol, ICF
Time Frame: Protocol and consent form will be available once approval is received from the research ethical board and will remain available.
Access Criteria: Access criteria will be specified in the plan for data sharing, once available.

REFERENCES:
- [Background] Gafar F, Yunivita V, Fregonese F, Apriani L, Aarnoutse RE, Ruslami R, Menzies D. Pharmacokinetics of standard versus high-dose rifampin for tuberculosis preventive treatment: A sub-study of the 2R2 randomized controlled trial. Int J Antimicrob Agents. 2024 Jul;64(1):107197. doi: 10.1016/j.ijantimicag.2024.107197. Epub 2024 May 14. PMID 38750674
- [Result] Fregonese F, Apriani L, Barss L, Benedetti A, Cook V, Fisher D, Fox GJ, Johnston J, Long R, Nguyen TA, Nguyen VN, Ruslami R, Menzies D. High dose rifampin for 2 months vs standard dose rifampin for 4 months, to treat TB infection: Protocol of a 3-arm randomized trial (2R2). PLoS One. 2023 Feb 2;18(2):e0278087. doi: 10.1371/journal.pone.0278087. eCollection 2023. PMID 36730240